CLINICAL TRIAL: NCT06951438
Title: STI Self-swab Testing At the Time of Telemed Medication Abortion Provision
Brief Title: Assessing Acceptability and Feasibiity of STI Self-swab Testing, to be Offered at the Time of Telemed Medication Abortion Provision
Acronym: STAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: University of Hawaii Foundation (Unknown)
Responsible Party: Principal Investigator, Olivia Manayan, MD MPH, Principal Investigator, Queen's Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RA-2025-009
Record Dates: First submitted 2025-03-18; First posted 2025-04-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Sexually Transmitted Disease (STD); Gonorrhea; Chlamydia; Trichomonas Infection
Keywords: STI testing; telemedicine; medication abortion; self-swab collection; vaginal swab
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections; Trichomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Self-swab Arm (Experimental): These patients will be recruited to the study actively. Upon signing an informed consent, they will be instructed to collect an at-home, self-swab test for STI testing. The kit for collection will be provided for them, as well as the shipping materials for the specimen.
  Interventions: Diagnostic Test: Self-swab collection PCR test for chlamydia, gonorrhea, trichomonas
- in-clinic STI testing arm (No Intervention): This population will not be actively recruited. Demographic data will be collected for comparison to the intervention arm via retrospective chart review of a contemporaneous, in-clinic population seeking abortion care.

INTERVENTIONS:
Diagnostic Test: Self-swab collection PCR test for chlamydia, gonorrhea, trichomonas — Self-swab collection PCR test for chlamydia, gonorrhea, trichomonas
  Arms: Self-swab Arm

SUMMARY:
The goal of this interventional study is to provide more access to STI testing for patients who seek abortion care through telemedicine, particularly for those whose access to STI testing is otherwise limited. The main questions it aims to answer are:

What is the acceptability, feasibility, and utilization of self-collected STI screening at the time of telemedicine medication abortion provision?

How does the uptake of such a service among patients receiving telemedicine abortion care compare to the population of patients who seek in-person medication abortion care?

What are the positivity rates for STIs in among patients receiving telemedicine medication abortion care compared to the positivity rates for a contemporaneous, in-clinic population?

What is the average time to between testing and treatment for patients who test positive for an STI using the self-collection service?

Researchers will compare the intervention group to a contemporaneous, in-clinic population on uptake of STI screening, as well as on positivity rates for the STIs tested.

Participants will be asked to perform self-swab collection for STI testing for gonorrhea, chlamydia, and trichomonas. They will be instructed to send their specimens to a lab using prepaid postage. Upon completion of sample collection and shipping, they will be asked to complete a survey assessing basic demographic information, as well as acceptability and feasibility of the intervention. Patients who test positive for an STI will be promptly provided/referred to treatment.

DETAILED DESCRIPTION:
Study Design:

This is an explorative cohort study that will assess the accessibility, feasibility, and utilization of a new intervention: at-home, self-collected STI testing at the time of medication abortion received through telemedicine services.

The study will take place within the Complex Family Planning clinic, the Options Center in Honolulu, Hawaii.

The intervention group will be recruited from the telemedicine medication abortion patients.

This group will be compared to the control group with data pulled from a chart review of a comparison cohort of patients seen for in-clinic medication abortion during a contemporaneous period.

Patients in the telehealth group may be physically based on any of the Hawaiian Islands but must have internet access for telehealth services. During the initial telemedicine consultation for medication abortion, the patient will be screened for eligibility using the eligibility criteria described as detailed below. If a patient is eligible for the study, they will be asked if they would like to be enrolled in the study in order to perform STI testing via self-collection. If they do not wish to participate in the study, resources for alternative ways to get STI testing will be provided to them.

If the patient expresses interest in the study, at the conclusion of their telemedicine visit for abortion care, they will redirected to a separate telemedicine visit with the research coordinator. The research coordinator will describe the study in further detail and obtain informed consent if the patient still wishes to proceed. Patients will sign consent forms via Adobe e-sign, a secure digital platform.

Once informed consent has been obtained, the research associate will do a short teaching session that reviews the following points with participants:

1. Contents of the specimen collection kit, which will include written instructions for specimen collection
2. How to collect the specimen (this may be done with illustrative models or drawings) and how to handle the specimen once it has been collected. This will include instructions on how to place the swab in the collection tube containing buffer solution, and how to send the swab to the lab. Patients will be instructed to collect their specimens for STI testing prior to taking their medications for medication abortion, in order to improve the ease of collection.
3. Verifying that patients are willing to receive a survey following specimen receipt via text message, and that they have a working mobile phone number.
4. Verifying that they accept receiving positive test results by phone.
5. Asking if, and how, patients would like to be notified of negative test results.

Patient information will be de-identified and connected to a unique Study ID. This study ID will label all specimens that patients send in the mail. All identifiable information, including signed consent forms, will be stored in a password protected and encrypted computer in the PI's research office on site.

The specimen collection kit will be included within the medication abortion kits, which are mailed to patients using a USPS bubble mailer. The patients will be able to locate their package by using a USPS tracking number once the kits have been mailed to them. Within the mailer, collection instructions and a prepaid envelope to send the specimens for processing will also be included. No PHI will be included in the specimen collection kit; all study materials sent to the laboratory for processing will be labeled only with the patient's study ID number.

Once the medication abortion kit and swab collection kit have been received, patients will perform self-swab collection before they initiate their medication abortion and send their specimen to the processing lab using the prepaid envelope provided for them. All specimens will be processed at the Emory Clinical Labs in Atlanta, GA. Once the lab has confirmed specimen receipt, the participant will receive a link via text message or email from the study team at QMC to a survey that assesses the acceptability and feasibility of the self-swab. This is a modified version of a validated survey that is used assess acceptability feasibility of telehealth-based interventions.18 The survey will also collect limited and non-identifiable demographic information. There will be a free-text portion at the end for patients to input any additional feedback regarding the intervention.

Once STI tests have been processed, the results will be emailed back to the research team using secure QMC email. All results sent through email will be deidentified, using only the patient's study ID number to identify the results. The lab staff will notify the PI if a submitted specimen is deemed inadequate for processing. If the swab is deemed inadequate, the research team will offer the patient the opportunity to swab again and provide them with a new test kit. Once the research team has received the results, they will be reported to the patient and scanned into the patient's electronic medical record.

If the lab staff does not receive a specimen from the patient prior to the patient's scheduled medication abortion follow-up appointment (typically scheduled 1-2 weeks after the initial consultation), the participant will be asked during the follow-up visit if they still desire or intend to send in a specimen, and reminded of the self-swab instructions if they express an intention to still complete the testing. If the patient does not attend her scheduled follow-up visit, one attempt will be made to contact her regarding specimen collection on the day of the scheduled appointment via phone call. If the study team is unsuccessful in contacting the patient at this time, no further attempts at contact will be made.

All patients who have a positive test result will be notified and provided options for treatment as soon as the research team is notified of the result. Patients may opt to receive negative test results via phone call (with option to approve leaving a detailed message on voicemail or not), Epic MyChart or text message, or opt out of receiving updates about negative test results.

Study population:

The study population will be patients living in Hawai'i who seek abortion care via telemedicine. The investigator team currently sees patients through telemedicine on six of the Hawaiian Islands (O'ahu, Maui, Hawai'i island, Kaua'i, Moloka'i, and Lāna'i). For many patients, specifically those located on Kaua'i, Lāna'i, and Moloka'i, medication abortion is the only option available for termination without having to fly to see an abortion provider. While Kaua'i has several in-person providers who provide medication abortion, on Lāna'i and Moloka'i, there are no providers on island who provide medication abortions in clinic, so telemedicine medication abortion is their only option.

Number of subjects

The investigator team will enroll a total of 75 subjects for this study. The guidance for determining sample sizes in pilot studies assessing feasibility recommends 70-100 subjects, which will allow analysis for correlation between variables without sacrificing significant confidence intervals. Additionally, in a very similar feasibility study assessing a telehealth STI intervention for same-sex male couples,15 the sample comprised of 50 couples, with samples collected from 100 study subjects.

For the contemporaneous, in-clinic population that will serve as the control group, all charts for patients who receive medication abortion in the same time frame that recruitment for the study took place will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of the Queen Medical Center Options Center clinic seeking telemedicine medication abortion.
2. Patients for whom, according to the CDC guidelines for STI Testing11, STI testing is indicated, or patients who desire STI screening
3. Age 14 and over
4. Can speak and read English
5. Displays capacity for informed consent

Exclusion Criteria:

1. Home address that is not located in the state of Hawai'i
2. Incarcerated
3. Unwilling to perform vaginal swab collection

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants must be pregnant in order to participate
Enrollment: 75 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Utilization of self-collected STI screening at the time of telemedicine medication abortion provision | 1) up to one year 2) up to one year
  Utilization rates will be reported as a percentage. Both enrollment in the study, as well as utilization of the actual STI testing services, will be reported as measures of utilization. The former (1) will be reported as the percentage of eligible patients who chose to enroll in the study, while the latter (2) will be reported as the percentage of enrolled patients who submitted samples for STI testing.
Acceptability of self-collected STI screening at the time of telemedicine medication abortion provision | Up to two weeks after completion of the intervention
  Acceptability will be measured using a modified version of the Digital Health Acceptability Questionnaire (DHAQ) which is a validated survey that is used to assess acceptability and feasibility of telehealth-based interventions. The first five questions (1-5) are validated to assess attitude toward the service as a means to address healthcare needs, while the second five questions (6-10) address individual capacity and effort to use the telehealth intervention. A copy of this survey can be found in Table A. This is a 10 question survey of Likert scales from 1 to 5, with 1 being "Strongly Disagree" and 5 being "Strongly Agree".
  We will calculate median and IQR across the domains of the DHAQ to determine a median acceptability score, which will be calculated using the scores from questions 1-5.
Feasibility of self-collected STI screening at the time of telemedicine medication abortion provision | 1) Up to two weeks after completion of the intervention
  Feasibility will be measured using a modified version of the Digital Health Acceptability Questionnaire (DHAQ) which is a validated survey that is used to assess acceptability and feasibility of telehealth-based interventions. The first five questions (1-5) are validated to assess attitude toward the service as a means to address healthcare needs, while the second five questions (6-10) address individual capacity and effort to use the telehealth intervention. A copy of this survey can be found in Table A. This is a 10 question survey of Likert scales from 1 to 5, with 1 being "Strongly Disagree" and 5 being "Strongly Agree".
  We will calculate median and IQR across the domains of the DHAQ to determine a median acceptability score, which will be calculated using the scores from questions 6-10.

SECONDARY OUTCOMES:
Comparison of uptake and STI positivity rates between the telehealth and in-clinic population | up to one year
  Once enrollment is complete for the telemedicine patient-recruitment, we will conduct a chart review of contemporaneous patients seen in-clinic for medication abortion, assessing for the percentage of patients who were offered and accepted STI testing, as well as for the positivity rates of chlamydia, gonorrhea, and trichomonas in this population.
Time elapsed between test result and prescription for treatment for patients who have a positive test for STI | one week
  For every patient who tests positive for an STI, we will measure the amount of time it takes from the time the patient is notified of their positive test result until the time the patient is sent treatment in the mail (chlamydia), or until a prescription for treatment is sent to the patient's pharmacy of choice (gonorrhea or trichomonas). The times will be reported as a range, as well as analyzed using measures of central tendency.

CONTACTS AND LOCATIONS:
Locations (1):
- Queens Medical Center, 1004 Clinic POB1, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will be anonymized.

REFERENCES:
- [Background] Gaydos CA, Cartwright CP, Colaninno P, Welsch J, Holden J, Ho SY, Webb EM, Anderson C, Bertuzis R, Zhang L, Miller T, Leckie G, Abravaya K, Robinson J. Performance of the Abbott RealTime CT/NG for detection of Chlamydia trachomatis and Neisseria gonorrhoeae. J Clin Microbiol. 2010 Sep;48(9):3236-43. doi: 10.1128/JCM.01019-10. Epub 2010 Jul 28. PMID 20668135
- [Background] US Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for HIV, STD and TB Prevention (NCHSTP), Division of STD/HIV Prevention, Sexually Transmitted Disease Morbidity for selected STDs by age, race/ethnicity and gender 1996-2014, CDC WONDER Online Database. Accessed 2025 Jan 7. http://wonder.cdc.gov/std-race-age.html.
- [Background] The Guttmacher Institute. State laws and policies: An overview of consent to reproductive health services by young people. Published 2023 Aug 30. Accessed 2024 Dec 26. https://www.guttmacher.org/state-policy/explore/overview-minors-consent-law
- [Background] Committee Opinion No. 665: Guidelines for Adolescent Health Research. Obstet Gynecol. 2016 Jun;127(6):e183-e186. doi: 10.1097/AOG.0000000000001486. PMID 27214193
- [Background] Haydon HM, Major T, Kelly JT, Catapan SC, Caffery LJ, Smith AC, Gallegos-Rejas V, Thomas EE, Banbury A, Snoswell CL. Development and validation of the Digital Health Acceptability Questionnaire. J Telemed Telecare. 2023 Dec;29(10_suppl):8S-15S. doi: 10.1177/1357633X231202279. PMID 38007698
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Spielberg F, Levy V, Lensing S, Chattopadhyay I, Venkatasubramanian L, Acevedo N, Wolff P, Callabresi D, Philip S, Lopez TP, Padian N, Blake DR, Gaydos CA. Fully integrated e-services for prevention, diagnosis, and treatment of sexually transmitted infections: results of a 4-county study in California. Am J Public Health. 2014 Dec;104(12):2313-20. doi: 10.2105/AJPH.2014.302302. Epub 2014 Oct 16. PMID 25320878
- [Background] Sullivan SP, Sullivan PS, Stephenson R. Acceptability and Feasibility of a Telehealth Intervention for STI Testing Among Male Couples. AIDS Behav. 2021 Dec;25(12):4029-4043. doi: 10.1007/s10461-021-03173-4. Epub 2021 Jan 28. PMID 33507455
- [Background] Lunny C, Taylor D, Hoang L, Wong T, Gilbert M, Lester R, Krajden M, Ogilvie G. Self-Collected versus Clinician-Collected Sampling for Chlamydia and Gonorrhea Screening: A Systemic Review and Meta-Analysis. PLoS One. 2015 Jul 13;10(7):e0132776. doi: 10.1371/journal.pone.0132776. eCollection 2015. PMID 26168051
- [Background] Center for Disease Control. Screening recommendations and considerations referenced in treatment guidelines and original sources. Published 2024 Mar 22. Accessed 2024 Oct 1. https://www.cdc.gov/std/treatment-guidelines/screening-recommendations.htm
- [Background] Norris A, Upadhyay U, O'Donnell J, et al. #WeCount report: April 2022 to June 2024. Society of Family Planning. Published 2024 Oct 22. doi:10.46621/728122kflzwf
- [Background] Kerestes C, Murayama S, Tyson J, Natavio M, Seamon E, Raidoo S, Lacar L, Bowen E, Soon R, Platais I, Kaneshiro B, Stowers P. Provision of medication abortion in Hawai'i during COVID-19: Practical experience with multiple care delivery models. Contraception. 2021 Jul;104(1):49-53. doi: 10.1016/j.contraception.2021.03.025. Epub 2021 Mar 28. PMID 33789080
- [Background] Barrow RY, Ahmed F, Bolan GA, Workowski KA. Recommendations for Providing Quality Sexually Transmitted Diseases Clinical Services, 2020. MMWR Recomm Rep. 2020 Jan 3;68(5):1-20. doi: 10.15585/mmwr.rr6805a1. PMID 31899459
- [Background] McNicholas C, Madden T, Secura G, Peipert JF. The contraceptive CHOICE project round up: what we did and what we learned. Clin Obstet Gynecol. 2014 Dec;57(4):635-43. doi: 10.1097/GRF.0000000000000070. PMID 25286295
- [Background] Frost JJ, Gold RB, Bucek A. Specialized family planning clinics in the United States: why women choose them and their role in meeting women's health care needs. Womens Health Issues. 2012 Nov-Dec;22(6):e519-25. doi: 10.1016/j.whi.2012.09.002. PMID 23122212
- [Background] Frost JJ, Mueller J, Pleasure ZH. Trends and differentials in receipt of sexual and reproductive health services in the United States: services received and sources of care, 2006-2019. Guttmacher Institute. https://www.guttmacher.org/report/sexual-reproductive-health-services-in-us-sources-care-2006-2019. Published 2021 Jun.
- [Background] Srinivas M, Wong NS, Wallace R, Emch M, Tang W, Yang EJ, Tucker JD. Sexually Transmitted Infection Rates and Closure of Family Planning Clinics Because of Abortion Restrictions in Iowa. JAMA Netw Open. 2022 Oct 3;5(10):e2239063. doi: 10.1001/jamanetworkopen.2022.39063. PMID 36239943
- [Background] Baden K, Dreweke J, Gibson C. Clear and growing evidence that Dobbs is harming reproductive health and freedom. Published 2024 Aug 22. Accessed 2024 Oct 1. https://www.guttmacher.org/2024/05/clear-and-growing-evidence-dobbs-harming-reproductive-health-and-freedom.
- [Background] Abortion in the United States. Published 2024 Jun 25. Accessed 2024 Oct 1. https://www.guttmacher.org/fact-sheet/induced-abortion-united-states.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT06951438/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT06951438/ICF_001.pdf